CLINICAL TRIAL: NCT00607581
Title: An Open-label, Phase II Study of Cyclophosphamide, Lenalidomide and Dexamethasone (CLD) for Previously Treated Patients With AL Amyloidosis
Brief Title: Cyclophosphamide, Lenalidomide and Dexamethasone (CLD) for Previously Treated Patients With AL Amyloidosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Principal Investigator, Giampaolo Merlini, Director, Amyloidosis Treatment and Research Center, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AC-003-IT; RV-AMYL-PI-303
Record Dates: First submitted 2008-01-22; First posted 2008-02-05 (Estimated); Last update posted 2012-02-10 (Estimated); Status verified 2012-02

CONDITIONS: Amyloidosis
Keywords: amyloidosis; lenalidomide; cyclophosphamide; dexamethasone
MeSH Terms: conditions — Amyloidosis | interventions — Cyclophosphamide; Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): The participants receive up to 9 28-day cycles of
  * cyclophosphamide: 500 mg orally on days 1, 8, 15;
  * lenalidomide: 15 mg orally on days 1-21;
  * dexamethasone: 40 mg orally on days on days 1, 8, 15, 22.
  Interventions: Drug: cyclophosphamide; Drug: lenalidomide; Drug: dexamethasone

INTERVENTIONS:
Drug: cyclophosphamide — cyclophosphamide: 500 mg orally on days 1, 8, 15
  Other Names: Endoxan; D003520
Drug: lenalidomide — lenalidomide: 15 mg orally on days 1-21
  Other Names: Revlimid; CC 5013; C467567
Drug: dexamethasone — dexamethasone: 40 mg orally on days on days 1, 8, 15, 22
  Other Names: Soldesam; D003907

SUMMARY:
The treatment of light-chain (AL) amyloidosis is directed against the plasma cells that produce the light-chain forming the amyloid deposits. The plasma cells can be killed and their growth can be stopped by drugs used in chemotherapy, such as cyclophosphamide, steroids, such as dexamethasone, and drugs that stimulate the immune system, such as lenalidomide.

The present trial studies the efficacy and safety of the combination of cyclophosphamide, lenalidomide and dexamethasone in patients with AL amyloidosis who were previously treated and need further therapy.

DETAILED DESCRIPTION:
This study will include previously treated patients with AL amyloidosis.

Primary objectives to determine the hematologic and organ response rate to the association of cyclophosphamide, lenalidomide and dexamethasone (CLD).

Secondary objectives

* to determine the safety of CLD,
* to determine time to response to CLD,
* to determine the duration of response to CLD,
* to assess survival of AL amyloidosis patients treated with CLD.

Patients receive 28-day cycles cyclophosphamide on days 1, 8 and 15, oral lenalidomide on days 1-21 and oral dexamethasone on days 1, 8, 15, and 22.

Up to 9 courses can be performed until one of the following endpoints is met:

* completion of cycle 9,
* complete hematologic remission observed after cycle 3 or 6,
* partial hematologic response associated with organ response after cycle 6.
* no response at cycle 3 or 6. After completion of study treatment, patients are followed every 3 months for up to 3 years.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of AL amyloidosis.
* Evidence of a monoclonal light chain at serum and/or urine immunofixation electrophoresis.
* Elevated circulating free light chain (of the type identified by immunofixation) above the upper limit of the normal range and abnormal kappa/lambda ratio.
* Previously treated and requiring further treatment.
* Symptomatic organ involvement.
* Bone marrow plasma cell <30%.
* Echocardiographic ejection fraction >40%.
* Troponin I <0.1 ng/mL.
* Hemoglobin >10 g/dL.
* Absolute neutrophil count >1500/uL.
* Platelet count >140000/uL.
* Total bilirubin <2.5 mg/dL.
* Alkaline phosphatase <4 x upper reference limit (u.r.l.).
* ALT <3 x u.r.l..
* Glomerular filtration rate >30 mL/min.
* Performance status ECOG 1-3.
* Female subjects of childbearing potential must have two negative pregnancy tests prior to starting study drug.

Exclusion Criteria:

* Prior treatment with the association of cyclophosphamide, lenalidomide and dexamethasone or with lenalidomide.
* Requirement for other concomitant chemotherapy, immunotherapy or radiotherapy, or any investigational ancillary therapy.
* Presence of other active malignancies, with the exception of nonmelanoma skin cancer, cervical cancer, treated early-stage prostate cancer provided that prostate specific antigen is within normal limits.
* Clinically overt multiple myeloma.
* Uncontrolled infection.
* New York Heart Association (NYHA) class 4 heart failure.
* Enzyme documented myocardial infarction within 6 months before enrollment.
* Grade 2 or 3 atrioventricular block (Mobitz type I is permitted).
* Repetitive ventricular arrhythmias at 24 h Holter electrocardiogram in spite of treatment with amiodarone.
* Supine systolic blood pressure <90 mmHg, or symptomatic orthostatic hypotension, or a decrease in systolic blood pressure on standing of >20 mmHg in spite of being treated for orthostatic hypotension.
* Prior history of thrombosis or venous thromboembolism or pulmonary embolism. Prior diagnosis of antiphospholipid antibodies or lupus anticoagulant, factor V Leiden mutation, prothrombin G21210A mutation, antithrombin, protein C or S deficiency.
* Indication to receive clopidogrel, ticlopidine or warfarin.
* Factor X level <20%.
* Poorly controlled diabetes mellitus (if receiving antidiabetic agents, subjects must be on a stable dose for at least 3 months).
* Previous or ongoing psychiatric illness (with the exclusion of reactive depression).
* Pregnant or nursing women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2008-02; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
hematologic response rate | at 3 months

SECONDARY OUTCOMES:
organ response rate | at 3 months
time to response | every 28 days
time to progression | every 3 months for 3 years
survival | up to 3 years after treatment discontinuation
toxicity | continuous during treatment

CONTACTS AND LOCATIONS:
Overall Officials: Giampaolo Merlini, M.D., Principal Investigator — Fondazione IRCCS Policlinico San Matteo
Locations (1):
- Amyloidosis Research and Treatment Center - Fondazione IRCCS Policlinico San Matteo, Pavia, Pavia, Italy

REFERENCES:
- [Background] Wechalekar AD, Goodman HJ, Lachmann HJ, Offer M, Hawkins PN, Gillmore JD. Safety and efficacy of risk-adapted cyclophosphamide, thalidomide, and dexamethasone in systemic AL amyloidosis. Blood. 2007 Jan 15;109(2):457-64. doi: 10.1182/blood-2006-07-035352. Epub 2006 Sep 21. PMID 16990593
- [Background] Palladini G, Perfetti V, Perlini S, Obici L, Lavatelli F, Caccialanza R, Invernizzi R, Comotti B, Merlini G. The combination of thalidomide and intermediate-dose dexamethasone is an effective but toxic treatment for patients with primary amyloidosis (AL). Blood. 2005 Apr 1;105(7):2949-51. doi: 10.1182/blood-2004-08-3231. Epub 2004 Nov 30. PMID 15572585
- [Background] Dispenzieri A, Lacy MQ, Zeldenrust SR, Hayman SR, Kumar SK, Geyer SM, Lust JA, Allred JB, Witzig TE, Rajkumar SV, Greipp PR, Russell SJ, Kabat B, Gertz MA. The activity of lenalidomide with or without dexamethasone in patients with primary systemic amyloidosis. Blood. 2007 Jan 15;109(2):465-70. doi: 10.1182/blood-2006-07-032987. Epub 2006 Sep 28. PMID 17008538
- [Background] Sanchorawala V, Wright DG, Rosenzweig M, Finn KT, Fennessey S, Zeldis JB, Skinner M, Seldin DC. Lenalidomide and dexamethasone in the treatment of AL amyloidosis: results of a phase 2 trial. Blood. 2007 Jan 15;109(2):492-6. doi: 10.1182/blood-2006-07-030544. Epub 2006 Sep 7. PMID 16960148
- [Background] Merlini G, Stone MJ. Dangerous small B-cell clones. Blood. 2006 Oct 15;108(8):2520-30. doi: 10.1182/blood-2006-03-001164. Epub 2006 Jun 22. PMID 16794250
- [Derived] Palladini G, Russo P, Milani P, Foli A, Lavatelli F, Nuvolone M, Perlini S, Merlini G. A phase II trial of cyclophosphamide, lenalidomide and dexamethasone in previously treated patients with AL amyloidosis. Haematologica. 2013 Mar;98(3):433-6. doi: 10.3324/haematol.2012.073593. Epub 2012 Sep 14. PMID 22983583